CLINICAL TRIAL: NCT05285215
Title: Integrated Psychological Program for Management of Postnatal Depression and Persistent Postpartum Pain After Childbirth: CODEPAD - II (Collaborative Outcomes of DEpression and Pain Associated With Delivery- II)
Brief Title: Integrated Psychological Program for Management of Postnatal Depression and Persistent Postpartum Pain After Childbirth
Acronym: CODEPAD-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Sng Ban Leong, Head of Department, Women's Anaesthesia, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSAINV21jun-0008
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated psychological program (IPP) group (Experimental): Patients are assigned to have mindfulness training and music listening before and after delivery. Video counselling will be offered if patient is found to have Edinburgh Postnatal Depression Scale (EPDS) equal to or more than 10. Questionnaires on psychological and pain assessments will be administered before and after delivery, with the final time point being 2 months after delivery.
  Interventions: Procedure: Integrated psychological program (IPP)
- Non- Integrated psychological program (IPP) group (No Intervention): Questionnaires on psychological and pain assessments will be administered before and after delivery, with the final time point being 2 months after delivery.

INTERVENTIONS:
Procedure: Integrated psychological program (IPP) — Patients will listen to the music for 30 minutes before delivery, and resume music listening once they are comfortable after delivery. Upon discharge, they will be asked to have music listening at least 30 minutes per day until 8 weeks postnatal survey.
  Mindfulness training via mobile application is administered before delivery. After delivery, they are asked to perform mindfulness training for 10 minutes daily, until last follow-up at 8 weeks post-delivery.
  Mobile electronic survey will be used to assess patients' EPDS scores fortnightly, until the last follow-up at week 8 post-delivery. If the EPDS scoring is found to be equal to or more than 10, video counselling and/or face-to-face consultation will be arranged.
  Video counselling sessions will be offered if patients are found to have EPDS score of 10-12. For women found to have EPDS≥13, a face-to-face initial psychiatry consultation will be conducted.
  Arms: Integrated psychological program (IPP) group

SUMMARY:
The integrated psychological program (IPP) is based on evidence from the local population showing that the interventional components (mindfulness training, music listening, video counselling) are amenable to implementation in the outpatient care setting. Incorporating innovative digital mobile and electronic applications in the care of an increasingly technology-savvy population will be strategic. The proposal will transform the healthcare model for treating postnatal depression (PND) and persistent postpartum pain (PPP).

DETAILED DESCRIPTION:
The childbirth process is associated with the risk of developing postnatal depression (PND) and persistent postpartum pain (PPP), which could contribute to maternal morbidity. There is a lack of routine structured and effective programs in current practice to monitor and effectively manage PND and PPP. Pilot study found specific pain and psychological vulnerability factors associated with increased risk of PND after childbirth.

The investigators propose an integrated psychological program (IPP) consisting of mindfulness mobile application, music listening, digital health video counselling and mobile electronic survey to effectively prevent, detect, monitor, and treat PND and PPP. The primary aim is to determine whether the use of the IPP will result in lower incidence of PND after childbirth. The study will also determine whether the use of the IPP will result in lower postnatal Edinburgh Postnatal Depression Scale (EPDS) scores in a subgroup of laboring women (with outcomes of vaginal or emergency Cesarean delivery) that may have increased risk factors for PND. The interplay of psychological and pain factors during the use of the IPP will also be determined using patient centric outcomes (mother-child bonding, breastfeeding self-efficacy, quality of life). A total of 1480 women undergoing childbirth will be recruited in this randomized controlled trial.

This proposal has the potential to recommend guidelines in community care and to incorporate digital health in management of PND and PPP. The IPP will also provide patient-centered care tailored to the individual's needs and will have an immediate potential to improve transition of hospital to community care in postnatal women health.

ELIGIBILITY:
Inclusion Criteria:

* healthy (American Society of Anesthesiologists physical status 2)
* parturient women at term (36 weeks' gestation or more, nulliparous and multiparous);
* with a singleton fetus;
* to have delivery in this institution.

Exclusion Criteria:

* current active psychiatric care;
* history of intravenous drug or opioid abuse;
* previous history of chronic pain syndrome.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant patients giving birth in the institution will be recruited.
Enrollment: 1480 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postnatal depression in both groups | 8 weeks after delivery (2 months)
  Incidence of postnatal depression will be assessed via Edinburgh Postnatal Depression Scale (EPDS) score at week 8 after delivery. EPDS is a 10-item self reporting scale to evaluate the postnatal depression. Participants are asked to respond according to how they have felt in the past seven days. Each item is measured on a 4-point scale (0-3), with a total score in the range of 0 to 30. A higher total score indicates a greater degree of depressive symptoms. A score of 10 and above indicates clinically significant depressive symptoms.
The incidence of persistent postpartum pain (PPP) in both groups | 8 weeks after delivery (2 months)
  The incidence of PPP is defined as the presence of pain for 8 weeks at the perineal, surgical scar or abdominal region related to childbirth at week 8 after delivery.

SECONDARY OUTCOMES:
Breastfeeding self-efficacy in both groups | 8 weeks after delivery (2 months)
  The breastfeeding self-efficacy will be assessed by breastfeeding self-efficacy scale- short form (BSES-SF). Breastfeeding self-efficacy refers to a mother's confidence and perception of how well she can breastfeed her infant. The 14-item self-administered BSES-SF comes in a 5-point Likert-type scale where 1 indicates not at all confident and 5 indicates always confident. Scores are summed to produce a range from 14 to 70, with higher scores indicating higher levels of breastfeeding self-efficacy.
Postpartum bonding in both groups | 8 weeks after delivery (2 months)
  The postpartum bonding will be assessed by Postpartum Bonding Questionnaire (PBQ). It consists of 25 items on four sub scales: i) impaired bonding; ii) rejection and anger; iii) anxiety about care; and iv) risk of abuse. The items are based on Likert scale ranging from 0 (always) to 5 (never), with a total score ranging from 0 to 125 where lower PBQ scores are associated with better mother-child bonding.
Health status in both groups | 8 weeks after delivery (2 months)
  Health status will be assessed via EQ-5D-5L, a standardized instrument for measuring generic health status. It is made up for two components; health state description and evaluation. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each dimension ranging from 1-5 (5L). From these five dimensions, EQ-5D index is calculated, having a value between 0-1. The evaluation part involves an analogue scale, asking to mark health status on the day of the survey on a 20 cm vertical scale with end points of 0 and 100. Zero corresponds to " worst imaginable health state", and hundred corresponds to "best imaginable health state".

OTHER OUTCOMES:
Matching between intention and actual use of labor epidural analgesia | 1 day (during labor and delivery)
  Intention of the use of labor epidural analgesia (yes/ no/ not sure) will be asked and matched against the actual use of labor epidural analgesia (yes/ no) during labor and delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No